CLINICAL TRIAL: NCT05908981
Title: The Effects of Sandalwood Aromatherapy (Santalum Album) and Lavender Oil on Anxiety Levels of Pediatric Patients Undergoing Dental Extraction
Brief Title: The Effects of Sandalwood Aromatherapy on Anxiety Levels of Pediatric
Acronym: ESAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aisha Mohammed Hamzi (Other)
Collaborators: clinical professor (Unknown)
Responsible Party: Sponsor-Investigator, Aisha Mohammed Hamzi, The effects of sandalwood aromatherapy (Santalum album) and Lavender oil on anxiety levels of pediatric patients undergoing dental extraction., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: effects sandalwood on anxiety
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Anxiety, Dental
MeSH Terms: conditions — Anxiety Disorders | interventions — lavender oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effects of sandalwood oils on anxiety levels of pediatric (Active Comparator): first group sandalwood aromatherapy
  Interventions: Other: sandalwood aromatherapy (Santalum album)
- The effects of Lavender oils on anxiety levels of pediatric (Active Comparator): second group lavender oil
  Interventions: Other: sandalwood aromatherapy (Santalum album)

INTERVENTIONS:
Other: sandalwood aromatherapy (Santalum album) — Aromatherapy is a relaxation therapy media that uses aromatic essence extracts from plant parts. Aromatherapy is used to treat and improve physical and psychological health
  Other Names: Lavender oil

SUMMARY:
Aim of the study:

Evaluate the anxiety in the child before treatment. Detection of the sandalwood and lavender oil effect on dental anxiety.

DETAILED DESCRIPTION:
Anxiety is a kind of emotional disorder associated with unexpected or considered dangerous situations. Physiological signs that can be observed are sweating, increased blood pressure, tachycardia, dry mouth, diarrhea, muscle tension, and hyperventilation. The prevalence of anxiety for worldwide dental patients is considered high, reaching 6-15% of the population and usually starting from childhood (51%) and adolescents (22%). A study showed that 25% of primary-school-age children undergoing dental treatment experienced severe anxiety, 50% moderate anxiety, and 20% mild anxiety.

Aromatherapy is a relaxation therapy media that uses aromatic essence extracts from plant parts. Aromatherapy is used to treat and improve physical and psychological health. Aromatherapy essential oil stimulates receptors in the nose, then the information is transmitted further to areas in the brain that control emotions and provide information to the hypothalamus, which is a regulator of the internal system of the body so that it reacts to stress.

Sandalwood is one of 22 species of the genus Santalum in the world and is a commercial species through Santalol oil that is widely used as a feedstock for aromatherapy. Sandalwood has a distinctive aroma. This aroma comes from the main content of sandalwood, Santa lol. The quality of sandalwood oil is determined by the content of a-santalol and P-santalol. a-santalol and P-santalol are sesquiterpene organic compounds. Through aromatherapy, sandalwood oil is widely used to relieve anxiety, stress, and depression. This oil has neuroleptic, calming, and bronchial dilatation effects.

This study aims to analyze sandalwood aromatherapy's effect on the anxiety level of pediatric patients undergoing dental treatment. The analysis was seen through three indicators of anxiety, namely systolic blood pressure, diastolic blood pressure, and heart rate per minute.

ELIGIBILITY:
Inclusion Criteria:

1. Egyptian children from 6 to 12 years old undergo primary tooth extraction.
2. Absence of any systemic problems, physical and mental disabilities.
3. Children intellectually sufficient to complete the anxiety scale and those whose parents were willing to participate in the study.
4. Frankel rating 3 in cooperation.

Exclusion Criteria:

1. Presence of dental or medical emergency and systemic disorders.
2. Special needs children.
3. Children with any respiratory tract illnesses, common cold, or allergy.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
primary outcome it is pulse rate for child undergoing extraction | 3 month
  It is measurement by Automated pressure device ((unit of M blood minute (1-5)

SECONDARY OUTCOMES:
Secondary outcome anxiety level of anxiety and blood pressure | 3month
  measurement by Dental anxiety faces version ( MCDAS-simplified) scores from 1to 5 minimal it is 1 maximal it is 20 maximam it is wors Blood pressure measurement by Automated blood pressure device unit Millimetres of mercury

CONTACTS AND LOCATIONS:
Overall Officials: Kamal El-Motayam, Professor, Study Director — Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Mahendra, V. G., Dewi, A. M., Tedjosasongko, U., & Wibowo, T. B. (2020). The Effects of Sandalwood Aromatherapy (Santalum Album) and Bossa Nova Music on Anxiety Levels of Pediatric Patients Undergoing Topical Fluoride Treatment. European Journal of Molecular & Clinical Medicine, 7(5), 860-865.
- [Result] Lakhan SE, Sheafer H, Tepper D. The Effectiveness of Aromatherapy in Reducing Pain: A Systematic Review and Meta-Analysis. Pain Res Treat. 2016;2016:8158693. doi: 10.1155/2016/8158693. Epub 2016 Dec 14. PMID 28070420